CLINICAL TRIAL: NCT00001619
Title: Magnetic Resonance at 1.5 and 3 Tesla
Brief Title: Magnetic Resonance Imaging at Different Levels of Magnetic Intensity
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970026; 97-H-0026
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-20

CONDITIONS: Cardiovascular Disease; Healthy
Keywords: Imaging; Spectroscopy; MRI; Cardiovascular; Technical Development; Heart; Safety; Toxicity; Gadolinium; Adverse Events; Normal Volunteer
MeSH Terms: conditions — Cardiovascular Diseases

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic tool that creates high quality images of the human body without the use of X-ray (radiation). MRI uses different levels of magnetic fields to create images of the body and organs. Occasionally, researchers will give patients undergoing a MRI an injection of a substance called gadolinium. Gadolinium works by brightening areas of the magnetic resonance image, thereby improving the contrast.

In this study researchers will use magnetic resonance imaging and contrast substances, like gadolinium, on normal volunteers in order to evaluate different aspects of its performance. Information gathered from this study may be used to develop more specific research studies involving MRI.

DETAILED DESCRIPTION:
Technical evaluation of magnetic resonance imaging and spectroscopy will be performed on normal volunteers. These studies will be conducted in the MRI systems located at the NIH. These studies may involve the intravenous administration of commercially available MR contrast media and exercise. The results will be used to evaluate the performance of various pulse sequences, gradient coils, and RF coils on human subjects and will provide essential ground work for specific patient protocols.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any normal volunteer greater than or equal to 18 who is capable of giving informed consent.

EXCLUSION CRITERIA:

A subject will be excluded if he/she has a contraindication to MR scanning such as:

1. Brain aneurysm clip
2. Implanted neural stimulator
3. Implanted cardiac pacemaker or defibrillator
4. Cochlear or ear implant
5. Ocular foreign body (e.g. metal shavings)
6. Insulin pump
7. Pregnant women (when uncertain, subject will undergo urine or blood testing).
8. Claustrophobia
9. Any condition in the Principal Investigator's judgement which present unnecessary risk

EXCLUSION CRITERIA FOR GADOLINIUM ENHANCED STUDIES:

1. Lactating Women
2. Renal or hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 497 (Actual)
Dates: Start 1996-11-05; Study Completion 2011-07-20

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mattay VS, Weinberger DR, Barrios FA, Sobering GS, Kotrla KJ, van Gelderen P, Duyn JH, Sexton RH, Moonen CT, Frank JA. Brain mapping with functional MR imaging: comparison of gradient-echo--based exogenous and endogenous contrast techniques. Radiology. 1995 Mar;194(3):687-91. doi: 10.1148/radiology.194.3.7862963.
- [Background] Niendorf HP, Dinger JC, Haustein J, Cornelius I, Alhassan A, Clauss W. Tolerance data of Gd-DTPA: a review. Eur J Radiol. 1991 Jul-Aug;13(1):15-20. doi: 10.1016/0720-048x(91)90049-2. PMID 1889423
- [Background] Frank JA, Mattay VS, Duyn J, Sobering G, Barrios FA, Zigun J, Sexton R, Kwok P, Woo J, Moonen C, et al. Measurement of relative cerebral blood volume changes with visual stimulation by 'double-dose' gadopentetate-dimeglumine-enhanced dynamic magnetic resonance imaging. Invest Radiol. 1994 Jun;29 Suppl 2:S157-60. doi: 10.1097/00004424-199406001-00052. No abstract available. PMID 7928216